CLINICAL TRIAL: NCT02917798
Title: Evaluating an Alternative Clinical Genetics Cancer Care Delivery Model: A Pilot Study of Patient Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 16-919
Record Dates: First submitted 2016-09-22; First posted 2016-09-28 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Prostate Cancer; Pancreas Cancer
Keywords: Genetic Testing; 16-919
MeSH Terms: conditions — Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Genetic Testing in Ovarian ,Prostate or Pancreas Cancer: This study is a prospective single-arm study to examine how an alternative clinical genetics cancer care delivery model affects ovarian, prostate or pancreas cancer patients' cognitions, emotions, and behaviors. Participants will be contacted 1 week (+/- 1 week) (Assessment #2; and 3 months (+/- 2 weeks) (Assessment #3;) following the telephone post-test counseling session to complete the follow-up assessments. These assessments will measure psychological and behavioral study constructs.
  Interventions: Behavioral: Assessments

INTERVENTIONS:
Behavioral: Assessments

SUMMARY:
This study will evaluate patients' experiences with having gynecologic or prostate medical oncologists and surgeons offer them genetic testing, and having genetic counselors return the test results to patients over the telephone. This is different from the usual approach to genetic testing, where gynecologic or prostate medical oncologists and surgeons refer their patients to a genetic counselor in order to have these tests done, and the genetic counselors return the test results to the patient in person or over the telephone. The investigators will only be evaluating this alternative way of providing genetic testing to ovarian or prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* MSK patient age 18 years or older.
* Diagnosed with or presumed by physician to have prostate cancer, or pancreatic cancer and recommended to undergo, currently undergoing, or having undergone active surveillance. (Patients with invasive epithelial ovarian cancer, peritoneal cancer, or fallopian tube cancer, or pancreas cancer are no longer eligible for inclusion as of Amendment 9. Patients with advanced prostate cancer who have not participated in active surveillance are no longer eligible for inclusion as of Amendment 10)
* Deemed to be clinically appropriate for multiplex genetic testing by their physician.
* Agreed to receive clinical multiplex genetic testing from their physician.
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Exclusion Criteria:

* Patients who do not or will not receive their ongoing cancer care at MSK.
* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation.
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.
* For ovarian cancer patients only: patient insured by a payer that does not provide coverage for multiplex genetic testing as delivered in this protocol (e.g., Cigna, United Health Care, or Oxford, (because these payers require genetic counseling by a genetics professional prior to testing).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian, prostate or pancreas cancer who are considered appropriate for multiplex genetic testing by their MSK DMT physician.
Sampling Method: Non-Probability Sample
Enrollment: 1047 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
baseline to post-results change in distress levels | 2 years
  Change in distress levels (HADS-Anxiety) from Baseline to Assessments #2 and #3, measured as an effect size among participants who receive a pathogenic variant(s), no pathogenic variant(s), and variant(s) of uncertain significance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carlo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/